CLINICAL TRIAL: NCT01224366
Title: A 24-week, Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of Vildagliptin 50mg Bid as an add-on Therapy to Insulin, With or Without Metformin, in Patients With Type 2 Diabetes Mellitus.
Brief Title: Efficacy and Safety of Vildagliptin as add-on Therapy to Insulin in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLAF237A23135
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Add-on to insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: Vildagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin
  Arms: Vildagliptin
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the efficacy and safety of vildagliptin add-on therapy to reduce HbA1c in patients with T2DM inadequately controlled by insulin, with or without concurrent metformin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of T2DM
* On a stable dose of insulin as defined by the protocol
* On a stable does of metformin (if applicable) as defined by the protocol
* Age 18 to 80 years
* HbA1c of 7.5 to 11.0%
* Body Mass Index (BMI) 22 to 40 kg/m2

Exclusion Criteria:

* Type 1 diabetes
* Short-acting or rapid-acting insulin
* Pregnancy or lactation
* Evidence of serious diabetic complications
* Evidence of serious cardiovascular complications
* Laboratory value abnormalities as defined by the protocol
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
HbA1c reduction | 24 weeks

SECONDARY OUTCOMES:
HbA1c reduction in subpopulation treated with insulin and with metformin | 24 weeks
HbA1c reduction in subpopulation treated with insulin and without metformin | 24 weeks
Reduction in FPG (overall and subpopulations) | 24 weeks
Responder rates (overall and subpopulations) | 24 weeks
Incidence of hypoglycemia and severe hypoglycemia (overall and subpopulations) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (66):
- Australia (5):
  - Novartis Investigative Site, Box Hill
  - Novartis Investigative Site, Heidelberg Heights
  - Novartis Investigative Site, Parkville
  - Novartis Investigative Site #1, Wollongong
  - Novartis Investigative Site #2, Wollongong
- Belgium (5):
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, La Louvière
  - Novartis Investigative Site, Ronse
- Czechia (3):
  - Novartis Investigative Site #1, Ostrava
  - Novartis Investigative Site #2, Ostrava
  - Novartis Investigative Site #3, Ostrava
- Germany (15):
  - Novartis Investigative Site, Aßlar
  - Novartis Investigative Site, Bensheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Einbeck
  - Novartis Investigative Site #1, Hamburg
  - Novartis Investigative Site #2, Hamburg
  - Novartis Investigative Site #3, Hamburg
  - Novartis Investigative Site #4, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site #1, Kassel
  - Novartis Investigative Site #2, Kassel
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Saarlouis
  - Novartis Investigative Site, Schliemannstadt Neubukow
  - Novartis Investigative Site, Tübingen
- Guatemala (5):
  - Novartis Investigative Site #1, Guatemala City
  - Novartis Investigative Site #2, Guatemala City
  - Novartis Investigative Site #3, Guatemala City
  - Novartis Investigative Site #4, Guatemala City
  - Novartis Investigative Site #5, Guatemala City
- Hong Kong (2):
  - Novartis Investigative Site #1, Hong Kong
  - Novartis Investigative Site #2, Hong Kong
- Hungary (5):
  - Novartis Investigative Site #1, Budapest
  - Novartis Investigative Site #2, Budapest
  - Novartis Investigative Site, Dunaújváros
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Szeged
- India (10):
  - Novartis Investigative Site, Indore
  - Novartis Investigative Site, Jaipur
  - Novartis Investigative Site, Karnāl
  - Novartis Investigative Site #2, Mumbai
  - Novartis Investigative Site #1, Mumbia
  - Novartis Investigative Site #1, Nagpur
  - Novartis Investigative Site #2, Nagpur
  - Novartis Investigative Site, Nashik
  - Novartis Investigative Site #1, Trivandrum
  - Novartis Investigative Site #2, Trivandrum
- Romania (5):
  - Novartis Investigative Site, Alba Iulia
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site #1, Oradea
  - Novartis Investigative Site #2, Oradea
  - Novartis Investigative Site, Târgu Mureş
- Slovakia (8):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site #1, Bratislava
  - Novartis Investigative Site #2, Bratislava
  - Novartis Investigative Site #3, Bratislava
  - Novartis Investigative Site #1, Košice
  - Novartis Investigative Site #2, Košice
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Štúrovo
- United Kingdom (3):
  - Novartis Investigative Site, Carmarthen
  - Novartis Investigative Site #1, Glasgow
  - Novartis Investigative Site #2, Glasgow

REFERENCES:
- [Result] Kozlovski P, Foley J, Shao Q, Lukashevich V, Kothny W. Vildagliptin-insulin combination improves glycemic control in Asians with type 2 diabetes. World J Diabetes. 2013 Aug 15;4(4):151-6. doi: 10.4239/wjd.v4.i4.151. PMID 23961326